CLINICAL TRIAL: NCT04678180
Title: Randomized Clinical Study Evaluating the Treatment Outcome of Combined Virtual Tic Training in Children and Adolescents With a Chronic Tic Disorder
Brief Title: Treatment Outcome of Combined Virtual Tic Training in Children and Adolescents With a Chronic Tic Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Judith Becker Nissen, MD, PhD, senior researcher, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1-10-72-231-20
Record Dates: First submitted 2020-12-09; First posted 2020-12-21 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-02

CONDITIONS: Chronic Tic Disorder
Keywords: Habit reversal training; Exposure response prevention; Children and adolescents; virtual training
MeSH Terms: conditions — Tic Disorders

STUDY DESIGN:
Intervention Model Description: Group 1: a combination of treatment using virtual training (secure interactive video training) and training at the hospital. In total, nine sessions using a combined training of HRT and ERP
  Group 2: a combination of treatment using self-instructive videos and training at the hospital. In total, nine sessions using a combined training of HRT and ERP
Who Masked: Outcomes Assessor
Masking Description: The assessor of outcome was blinded to any previous evaluations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual tic training (Experimental): A combination of treatment using virtual tic training and training at the hospital. In total nine sessions using a combined training of HRT and ERP. In four of the nine sessions (session 3, 5, 6, 7) training is performed as a virtual training. All sessions last 60 minutes
  Interventions: Behavioral: Combined HRT and ERP
- Video tic training (Experimental): A combination of treatment using self-instructive videos and training at the hospital. In total nine sessions using a combined training of HRT and ERP. Four of the nine sessions are completed at the hospital (session 1 and 2 are combined 120 minutes, session 4: 60 minutes, session 8: 60 minutes and session 9: 60 minutes). For all sessions, self-instructive videos have been recorded instructing the child and their families how they should perform the training
  Interventions: Behavioral: Combined HRT and ERP

INTERVENTIONS:
Behavioral: Combined HRT and ERP — tic training using the principles of HRT and ERP as to reduce tic intensity

SUMMARY:
Tics are unwanted, repetitive movements or sounds that are either simple or complex in appearance. Tic disorders often have a huge impact on children's life. The investigators have previously shown a positive outcome of tic training combining habit reversal training (HRT) and exposure response prevention (ERP) either as an individual therapy or in a group setting. However, young people and families are often busy, and having to use a full day as to attend to tic training often is difficult both for the young person and their families. Therefore, the present study focuses on the clinical outcome of combining virtual training with training at the hospital

DETAILED DESCRIPTION:
Tics are unwanted, brief, repetitive, non-rhythmic movements or sounds that are classified as either simple or complex. Dependent on duration, tics are divided into transient tics and chronic tics. Tic disorders often have an early age of onset and may have a major impact on a young person's life. Treatment of a chronic tic disorder primarily comprises therapeutic intervention which consists of ERP (Exposure Response Prevention) and/or HRT (Habit Reversal Training).

The purpose of the project is to

* Evaluate the treatment outcome of combined video consultation/participating in training sessions at the hospital and of combined self-instructed video training/participating in training sessions at the hospital.
* Compare the treatment outcome of supplementary virtual consultation and supplementary video training via an app with a previous study on the treatment outcome of attending individual therapy (NISSEN, 2018) by means of benchmarking.
* In addition, expound on the significance of sensory modulation (sensitivity), not-just-right experience and the child's perception with regard to the severity of chronic tics and treatment outcome. Also, to investigate whether insight, sensitivity and the not-just-right experience change during treatment.
* As the app is newly developed in relation to the present study, the investigators wish to clarify the participants' evaluation of the app using a newly developed questionnaire (designed for this project). For comparison, a questionnaire has been designed for evaluating the applicability of the supplementary video sessions.

When patients are referred to the Tourette outpatient clinic, Aarhus University Hospital, Psychiatry, a comprehensive diagnostic assessment is carried out. The assessment is based on a modified version of the Schedule for affective disorders and schizophrenia for school-age children - present and lifetime version (K-SADS-PL). The K-SADS-PL information is used for confirming the primary diagnosis of chronic tics and for ensuring that none of the exclusion criteria have been met.

Inclusion criteria

The inclusion criteria are defined based on the ICD-10 diagnosis (International Classification of Diseases and Related Health Problems):

Chronic motor/vocal tics (DF95.1) Tourette syndrome (DF95.2), Age spectrum: 9-17 years old

Exclusion criteria

The exclusion criteria are defined as follows:

Patients with comorbidity such as mental retardation (IQ = 70 or less), psychosis, severe depression requiring treatment, suicidal behavior/threats or severe eating disorder.

Participated in tics training based on HRT/ERP treatment within the last six months.

Oral and written consent will be obtained from parents and children/adolescents (age 15 years and older).

The study will be an open, randomized controlled clinical study for children and adolescents with chronic tics disorders. The participants will be randomized using computer-generated randomization based on age and sex.

The participants will either be randomized for tics training with attendance combined with virtual training (group 1) or a combination of attendance and self-instructed training via videos on an app (group 2). Both settings are based on the "Niks til Tics" manual (NISSEN, 2018) that describes training in Habit Reversal Training (HRT) and Exposure Response Prevention (ERP) over nine sessions. Thus, two treatment groups will be set up:

Group 1 (treatment group 1) will consist of nine entire sessions (60 min each), but where four out of the nine sessions will be converted to video consultations. The content of the video consultations is comparable to the information and training the patients would have received if they attended at the clinic and which are defined in the "Niks til Tics" manual.

Group 2 (treatment group 2) will comprise five entire sessions (60 min) with clinic attendance, but where sessions 1 and 2 will be combined into one session with a duration of 120 min, session 4 will be held as usual with attendance after five weeks, session 8 will be held ten weeks after session 4, and session 9 will be held after two months. In addition, patients in group 2 will be given the opportunity to talk to the therapist on the phone. For the group 2 training sessions, an app has been developed for teaching patients the tics training method. A new app session will be released at each new treatment session, and the content of the app videos will follow the information and training, which the patients would have received if they had attended at the clinic and which are defined in the "Niks til Tics" manual.

All tic training sessions will be individual. The primary outcome goal includes the Yale Global Tics Severity Scale (YGTSS) in session 8. In order to follow the treatment, a parent report questionnaire and a self-report questionnaire will be used and evaluated in accordance with YGTSS (Golden standard). The questionnaires are based on Parent Tic Questionnaire (PTQ). Secondary outcome measures are Screen for Child Anxiety Related Emotional Disorders (SCARED), the Mood and Feelings Questionnaire (MFQ), Premonitory Urge Scale (PUTS), Beliefs About Tics Scale (BATS), NJR-C (not just right experiences), CATS (thoughts about experiences children may be exposed to), W-tc (worrying thoughts) and motivation questionnaire, and the parents are asked to fill in CBCL, BQ (general information) as well as a sensory profile (about hypersensitivity).

Statistical analyses The primary analysis will comprise a comparison of effect sizes within the treatment group, that is, an assessment of the reduction in tic intensity during the eight sessions. The difference in tic intensity between baseline and session 8 will be assessed at t-test. Effect sizes will be calculated by a ratio of the mean difference and the standard deviation of the difference between baseline and session 8 (SD diff). The confidence interval for effect sizes will be calculated using non-parametric bootstrap with 100 replications. At group sizes of 30 with an expected uniform YGTSS baseline of 25 (randomized) and with an expected SD of 6.2 (from a previous study (NISSEN 2018)), and a strength of 0.8 it should be possible to detect a decrease of point 3.4 (from baseline to session 8), which is statistically significant.

Responder level will be defined as a 25% reduction of the YGTSS total tics score.

The secondary analyses will study the reduction in tic intensity between the two treatment groups using unpaired t-test. At a group size of 30 and expected end YGTSS of 15 (SD 6.2) and strength of 0.80 (from a previous study (NISSEN 2018)), a difference of 4.6 between the two groups will be statistically significant.

Predictor analysis: baseline characteristics and baseline tic severity between the two groups will be compared using univariate Chi test for categorical variables and t-tests for continuous variables.

Tic severity will be assessed by independent raters.

Using benchmarking, the results of this treatment study will be compared with the results from a previous treatment study on HRT/ERP (NISSEN, 2018).

ELIGIBILITY:
Inclusion Criteria: based on ICD-10 diagnosen (International Classification of Diseases and Related Health Problems):

* Chronic motor/vocal tics (DF95.1)
* Tourettes syndrom (DF95.2)

Exclusion Criteria:

Comorbidity including

* Mental retardering
* Psychosis
* Severe depression
* Suicidal behavior
* Severe anorexia or
* If they have participated in tic training with HRT and/or ERP during the last 6 months

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change of baseline Yale Global Tic Severity Scale (YGTSS) at 16 weeks, 24 weeks, 40 weeks, 68 weeks | Baseline,16 weeks, 24 weeks, 40 weeks, 68 weeks
  YGTSS - a clinician-administered semi-structured interview including a checklist of all tics present in the past week. It covers five dimensions divided into ten items including the number, frequency, intensity, complexity and interference of motor and vocal tics. Furthermore, it includes a separate evaluation of the functional impairment. Measures the change in total tic score and functional impairment. Interval 0-100, high score means a worse outcome

SECONDARY OUTCOMES:
Change of baseline Premonitory Urge Scale (PUTS) 6 weeks, 16 weeks, 24 weeks, 40 weeks, 68 weeks | Baseline, 6 weeks, 16 weeks, 24 weeks, 40 weeks, 68 weeks
  PUTS is a short self-reporting scale with nine items. It measures the tic-related premonitory urge. Measures the change of baseline premonitory urge score at different end points. Interval 1-4, high score means a worse outcome
Change of baseline Beliefs About Tics Scale (BATS) at 6 weeks, 16 weeks, 24 weeks, 40 weeks, 68 weeks | Baseline, 6 weeks, 16 weeks, 24 weeks, 40 weeks, 68 weeks
  BATS is a self-reporting scale with 20 items developed to assess the different beliefs children and adolescent experience in relation to tic symptoms and to suppressing their tic symptoms. Measures the change of baseline premonitory urge score at different end points. Interval 1-4, high score means a worse outcome
Change of baseline Parent and child self-evaluating questionnaire at 16 weeks, 24 weeks, 40 weeks, 68 weeks | Baseline,16 weeks, 24 weeks, 40 weeks, 68 weeks
  Based on the PTQ a self-evaluating questionnaire have been developed for the children and their parents. Interval 1-4, high score means a worse outcome. The results will be compared to the golden standard YGTSS

OTHER OUTCOMES:
Change of baseline Screen for Child Anxiety Related Emotional Disorders (SCARED) at 6 weeks, 16 weeks, 24 weeks, 40 weeks, 68 weeks | Baseline, 6 weeks, 16 weeks, 24 weeks, 40 weeks, 68 weeks
  SCARED includes separate versions for parents and the child/adolescent. Using 41 items rated on a three-point scale, the questionnaire assesses the occurrence of anxiety symptoms based on DSM-IV. Interval 0-2, high score means worse outcome
Change of baseline Mood and Feelings Questionnaire (MFQ) at 6 weeks, 16 weeks, 24 weeks, 40 weeks, 68 weeks | Baseline, 6 weeks, 16 weeks, 24 weeks, 40 weeks, 68 weeks
  MFQ assesses the occurrence of depressive symptoms, using 13 items rated on a three-point scale. Interval 0-2, high score means worse outcome
Change of NJR-C (not just right) at 6 weeks, 16 weeks, 24 weeks, 40 weeks, 68 weeks | Baseline, 6 weeks, 16 weeks, 24 weeks, 40 weeks, 68 weeks
  NJR-C is a self-reporting questionnaire with 19 items. The questionnaire focuses on the not-just experiences that are often encountered in patients with tic disorders or OCD. Interval questions 1-10: 0-1, question 12: 1-4, questions 13-19: 1-7, high score means worse measure
Change of Children automatic thought scale (CATS) at 6 weeks, 16 weeks, 24 weeks, 40 weeks, 68 weeks | Baseline, 6 weeks, 16 weeks, 24 weeks, 40 weeks, 68 weeks
  CATS is a 40-item questionnaire focusing on children's negative self-statements across both internalizing and externalizing problems. Interval 0-4, high score means worse measure
Baseline Motivation of treatment questionnaire | Baseline
  Motivation of treatment questionnaire is a 15-item questionnaire evaluated on a four-point likert-scale. The questionnaire focusses on the motivation of the child to participate in the training,. Interval 0-2
Change of baseline Sensory profile at 6 weeks, 16 weeks, 24 weeks, 40 weeks, 68 weeks | Baseline, 6 weeks, 16 weeks, 24 weeks, 40 weeks, 68 weeks
  Sensory Profile is a collection of questionnaires for different age groups. The aim of the questionnaires is to assess children's responses to commonly occurring sensory events and to evaluate the ability to process the sensorimotor impressions. Interval 1-5

CONTACTS AND LOCATIONS:
Overall Officials: Judith Nissen, phd, Principal Investigator — Department of Child and Adolescent Psychiatry, Aarhus University Hospital, Denmark
Locations (1):
- Department of child and adolescent Psychiatry, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abramovitch A, Reese H, Woods DW, Peterson A, Deckersbach T, Piacentini J, Scahill L, Wilhelm S. Psychometric Properties of a Self-Report Instrument for the Assessment of Tic Severity in Adults With Tic Disorders. Behav Ther. 2015 Nov;46(6):786-96. doi: 10.1016/j.beth.2015.06.002. Epub 2015 Jun 18. PMID 26520221
- [Result] Andren P, Aspvall K, Fernandez de la Cruz L, Wiktor P, Romano S, Andersson E, Murphy T, Isomura K, Serlachius E, Mataix-Cols D. Therapist-guided and parent-guided internet-delivered behaviour therapy for paediatric Tourette's disorder: a pilot randomised controlled trial with long-term follow-up. BMJ Open. 2019 Feb 15;9(2):e024685. doi: 10.1136/bmjopen-2018-024685. PMID 30772854
- [Result] Birmaher B, Brent DA, Chiappetta L, Bridge J, Monga S, Baugher M. Psychometric properties of the Screen for Child Anxiety Related Emotional Disorders (SCARED): a replication study. J Am Acad Child Adolesc Psychiatry. 1999 Oct;38(10):1230-6. doi: 10.1097/00004583-199910000-00011. PMID 10517055
- [Result] Leckman JF, Riddle MA, Hardin MT, Ort SI, Swartz KL, Stevenson J, Cohen DJ. The Yale Global Tic Severity Scale: initial testing of a clinician-rated scale of tic severity. J Am Acad Child Adolesc Psychiatry. 1989 Jul;28(4):566-73. doi: 10.1097/00004583-198907000-00015. PMID 2768151
- [Result] Neal M, Cavanna AE. "Not just right experiences" in patients with Tourette syndrome: complex motor tics or compulsions? Psychiatry Res. 2013 Dec 15;210(2):559-63. doi: 10.1016/j.psychres.2013.06.033. Epub 2013 Jul 10. PMID 23850205
- [Result] Nissen JB, Kaergaard M, Laursen L, Parner E, Thomsen PH. Combined habit reversal training and exposure response prevention in a group setting compared to individual training: a randomized controlled clinical trial. Eur Child Adolesc Psychiatry. 2019 Jan;28(1):57-68. doi: 10.1007/s00787-018-1187-z. Epub 2018 Jun 28. PMID 29956034
- [Result] Ricketts EJ, Goetz AR, Capriotti MR, Bauer CC, Brei NG, Himle MB, Espil FM, Snorrason I, Ran D, Woods DW. A randomized waitlist-controlled pilot trial of voice over Internet protocol-delivered behavior therapy for youth with chronic tic disorders. J Telemed Telecare. 2016 Apr;22(3):153-62. doi: 10.1177/1357633X15593192. Epub 2015 Jul 13. PMID 26169350
- [Result] Singer HS. Tics and Tourette Syndrome. Continuum (Minneap Minn). 2019 Aug;25(4):936-958. doi: 10.1212/CON.0000000000000752. PMID 31356288
- [Result] Steinberg T, Harush A, Barnea M, Dar R, Piacentini J, Woods D, Shmuel-Baruch S, Apter A. Tic-related cognition, sensory phenomena, and anxiety in children and adolescents with Tourette syndrome. Compr Psychiatry. 2013 Jul;54(5):462-6. doi: 10.1016/j.comppsych.2012.12.012. Epub 2013 Jan 15. PMID 23332555
- [Result] Wood A, Kroll L, Moore A, Harrington R. Properties of the mood and feelings questionnaire in adolescent psychiatric outpatients: a research note. J Child Psychol Psychiatry. 1995 Feb;36(2):327-34. doi: 10.1111/j.1469-7610.1995.tb01828.x. PMID 7759594
- [Result] Woods DW, Piacentini J, Himle MB, Chang S. Premonitory Urge for Tics Scale (PUTS): initial psychometric results and examination of the premonitory urge phenomenon in youths with Tic disorders. J Dev Behav Pediatr. 2005 Dec;26(6):397-403. doi: 10.1097/00004703-200512000-00001. PMID 16344654
- [Result] ACHENBACH TM. Child behavior checklist and related instruments. In The use of psychological testing for treatment planning and outcome assessment. Edited by Maurish ME. Hillsdale, NJ: Lawrence Erlbaum Associates, 1994
- [Result] CHANG, S. Initial Psychometric Properties of a Brief Parent-Report Instrument for Assessing Tic Severity in Children with Chronic Tic Disorders. HIMLE, M. B.;TUCKER, B. T. P., et al. Child & Family Behavior Therapy: Taylor & Francis Group. 31: 181-191 p. 2009.
- [Result] Hedman E, Ljotsson B, Lindefors N. Cognitive behavior therapy via the Internet: a systematic review of applications, clinical efficacy and cost-effectiveness. Expert Rev Pharmacoecon Outcomes Res. 2012 Dec;12(6):745-64. doi: 10.1586/erp.12.67. PMID 23252357
- [Result] Martino D, Pringsheim TM. Tourette syndrome and other chronic tic disorders: an update on clinical management. Expert Rev Neurother. 2018 Feb;18(2):125-137. doi: 10.1080/14737175.2018.1413938. Epub 2017 Dec 8. PMID 29219631
- [Result] TEODORO M. Children's Automatic Thoughts Scale (Cats): adaptation and psychometric properties. Psico-USF [online], vol.18, n.1, pp.89-98. ISSN 1413-8271. https://doi.org/10.1590/S1413-8271201300100010, 2013